CLINICAL TRIAL: NCT04454112
Title: Pre and Post-gastrostomy Evaluation of Gastroesophageal Reflux in Children Using 24-hour pH Monitoring
Brief Title: Pre and Post-gastrostomy Evaluation of GER in Children Using 24-hour pH Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fatma Demirbaş (Other)
Responsible Party: Sponsor-Investigator, Fatma Demirbaş, Doctor of Pediatric Gastroenterology, Ondokuz Mayıs University
Organization: Ondokuz Mayıs University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2019/192
Record Dates: First submitted 2020-06-24; First posted 2020-07-01 (Actual); Last update posted 2020-07-01 (Actual); Status verified 2020-06

CONDITIONS: Gastroesophageal Reflux
MeSH Terms: conditions — Gastroesophageal Reflux

STUDY DESIGN:
Intervention Model Description: to compare the results of pre- and postoperative 24-hour pH monitoring in patients who underwent gastrostomy only and who underwent fundoplication concurrently with gastrostomy and to evaluate influence of gastrostomy/ LNF+ gastrostomy on GER.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- 24-hour esophageal pH monitoring (Experimental): 24-hour esophageal pH monitoring was conducted using an ambulatory system (Ohmega, MMS, Enschede, The Netherlands). This system consists of a portable data logger (MMS Investigation and Diagnostic Software®) and a disposable catheter which contains two pH electrodes (Unisensor, Attikon, Switzerland). Before recording, the pH electrode was calibrated in the special buffer solutions at pH values of 1 and 2.
  Interventions: Device: 24-hour esophageal pH monitoring using an ambulatory system (Ohmega, MMS, Enschede, The Netherlands).

INTERVENTIONS:
Device: 24-hour esophageal pH monitoring using an ambulatory system (Ohmega, MMS, Enschede, The Netherlands). — 24-hour esophageal pH monitoring application

SUMMARY:
The aim of this study was to evaluate 24-hour pH monitoring results before and after gastrostomy in neurological impaired (NI) children who underwent gastrostomy or Nissen fundoplication (NF) concurrently with gastrostomy.

DETAILED DESCRIPTION:
Gastrointestinal (GI) problems causing malnutrition may develop quite frequently in patients with neuromotor developmental delay. Diagnosis of GERD in patients with neurological impairment (NI) might be more difficult due to the absence of characteristic features in many cases. One of the best methods for the diagnosis of GER is the 24-hour esophageal pH monitoring.Even though there are some statements in the literature advocating that gastroesophageal reflux may develop in the late period in patients undergoing only gastrostomy, there are also reports supporting that gastrostomy does not contribute to the development of reflux.Regardless of whether the patient received anti-reflux surgery or not, the long-term follow-up is necessary in patients feeding with gastrostomy.The aim of this study is to compare the results of pre- and postoperative 24-hour pH monitoring in patients who underwent gastrostomy only and who underwent fundoplication concurrently with gastrostomy and to evaluate influence of gastrostomy/ LNF+ gastrostomy on GER.

ELIGIBILITY:
Inclusion Criteria:

Clinical diagnosis of neurological damage Must be able to apply gastrostomy or Nissen fundoplication concurrently with gastrostomy.

exclusion Criteria: to use anti-reflux medications long period of time gastroesophageal reflux disease

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2018-03-12 (Actual); Primary Completion 2018-12-12 (Actual); Study Completion 2018-12-12 (Actual)

PRIMARY OUTCOMES:
Pre and post-gastrostomy evaluation of gastroesophageal reflux in children using 24-hour pH monitoring | 2 month
  NI patients who had previously received pre and post-gastrostomy (Group 1) or gastrostomy+NF (Group 2) were underwent pH monitoring pre-post operatively.

SECONDARY OUTCOMES:
Pre and post-gastrostomy evaluation of gastroesophageal reflux in children using 24-hour pH monitoring | 7 month
  NI patients who had previously received pre and post-gastrostomy (Group 1) or gastrostomy+NF (Group 2) were underwent pH monitoring pre-post operatively.

CONTACTS AND LOCATIONS:
Overall Officials: Berat Dilek Demirel, Study Chair — she underwent gastrostomy to patients with neurological damage
Locations (1):
- Ondokuz Mayıs University Faculty of Medicine, Department of Pediatric Gastroenterology, Hepatology and Nutrition,, Kurupelit, Samsun, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No